CLINICAL TRIAL: NCT02833480
Title: A Study to Investigate the Differential Effects of Inhaled Symbicort and Advair on Lung Microbiota
Acronym: DISARM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Don Sin, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-02277
Record Dates: First submitted 2016-05-26; First posted 2016-07-14 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Budesonide, Formoterol Fumarate Drug Combination; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone group (Experimental): Advair (fluticasone) 250 mcg to be administered twice daily via Diskus for 12 weeks
  Interventions: Drug: Fluticasone group
- Budesonide group (Experimental): Symbicort (budesonide) 400 mcg to be administered twice daily via Turbuhaler for 12 weeks
  Interventions: Drug: Budesonide group
- Formoterol group (Active Comparator): Oxeze (formoterol) 12 microg to be administered twice daily via Turbuhaler for 12 weeks
  Interventions: Drug: Formoterol group

INTERVENTIONS:
Drug: Fluticasone group
  Other Names: Advair
  Arms: Fluticasone group
Drug: Budesonide group
  Other Names: Symbicort
  Arms: Budesonide group
Drug: Formoterol group
  Other Names: Oxeze
  Arms: Formoterol group

SUMMARY:
This study will evaluate the effects of budesonide (using Symbicort which is budesonide and formoterol) and fluticasone (using Advair which is fluticasone and salmeterol) on the airway microorganisms of patients with moderate-to-severe chronic obstructive pulmonary disease (COPD). This is a randomized, parallel group, two-centered clinical trial study to evaluate the effects of a 12 week treatment with Symbicort 400 mcg BID and Advair 250 mcg BID (via Diskus) on airway microbiota in patients with moderate-to-severe COPD. The control arm of this study will be Oxeze 12 ug BID.

DETAILED DESCRIPTION:
This is a randomized, non-placebo controlled study to evaluate the effects of Symbicort 400 mcg twice daily (BID) and Advair 250 mcg BID over 12 weeks. As the standard of therapy for COPD is a long-acting muscarinic antagonist (LAMA) treatment, a placebo only group cannot be ethically justified. The control arm of this study will thus be Oxeze 12 ug BID. The study will recruit approximately 69 subjects, from St. Paul's Hospital and British Columbia Cancer Agency, randomized 1:1:1 to the 3 arms in blocks. We anticipate 10 to 15% drop out rate, which will enable approximately 60 subjects for full analysis.

After the initial enrolment and confirmation of the entry criteria, subjects will perform spirometry before and following bronchodilation with salbutamol (up to 400 ug). They will then enter a 4-week run-in period during which all subjects will be withdrawn from inhaled corticosteroid containing products. They will then be treated with formoterol via Turbuhaler 12 ug BID and short-acting beta-2 agonists as needed (PRN). Subjects may also have LAMA (either tiotropium 18 ug once daily or glycopyrronium 50 ug once daily) at the discretion of the attending physician. At the end of the run-in phase, eligibility will be confirmed and then subjects will undergo pre and post-spirometry, low-dose thoracic computed tomography (CT) and bronchoscopy. One week post-bronchoscopy, the subjects will be randomized to a 12-week treatment period. Subjects may also have LAMA at the discretion of the attending physician. At the end of the 12 week treatment period, the subjects will undergo pre- and post-spirometry and 2nd bronchoscopy. The subjects will be re-evaluated one week following bronchoscopy and then discharged from the study. All subjects with pulmonary nodule requiring follow-up will be evaluated by the attending physician and the pulmonary nodule will be investigated as per guidelines of the Fleischner Society.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* History of moderate to very severe COPD with a post-bronchodilator forced expiratory volume/forced vital capacity (FEV1/FVC) <0.70 and a post-bronchodilator FEV1>20% and ≤80% of predicted normal value at screening.
* Current smoker or ex-smoker with a tobacco history of ≥10 pack-years (1 pack year= 20 cigarettes smoked per day for 1 year).

Exclusion Criteria:

* Clinically important pulmonary disease other than COPD (e.g. active lung infection, clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, and primary ciliary dyskinesia) and/ or radiological findings suggestive of a respiratory disease other than COPD that is contributing to the subject's respiratory symptoms.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

  1. Affect the safety of the subject throughout the study
  2. Influence the findings of the study or their interpretation
  3. Impede the subject's ability to complete the entire duration of study Subjects who have epilepsy must be on a stable dose of medication for 30 days prior to Visit 4.
* Unstable ischemic heart disease, or uncontrolled arrhythmia, cardiomyopathy, heart failure, and renal failure, or uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator
* Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 8 weeks prior to enrolment (Visit 1), based on last dose of steroids or last date of hospitalization whatever occurred later.
* Acute upper or lower respiratory infection requiring antibiotics or antiviral medication within 2 weeks prior to enrolment (Visit 1).
* Pneumonia within 8 weeks prior to enrolment (Visit 1), based on the last day of antibiotic treatment or hospitalization date, whatever occurred later.
* Pregnant, breastfeeding, or lactating women.
* Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening/run-in period, which, in the opinion of the Investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to complete entire duration of the study.
* Use of immunosuppressive medication, including rectal corticosteroids, high potency topical corticosteroids and systemic steroids within 28 days prior to randomization.
* Receipt of blood products within 30 days prior to enrollment (Visit 1).
* Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to Visit 1.
* History of alcohol or drug abuse within the past year, which may compromise the study data interpretation as judged by Investigator or Study Physician.
* Subjects who in the opinion of the investigator or qualified designee have evidence of active tuberculosis (TB), either treated or untreated.
* Scheduled in-patient hospitalization or surgical procedure during the course of the study.
* Asthma as a primary or main diagnosis according to the Global Initiative for Asthma (GINA, http://www.ginasthma.org/) guidelines or other accepted guidelines. Subjects with a past medical history of asthma (e.g. childhood or adolescence) may be included.
* The male partner of someone who may become pregnant during the course of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2015-02; Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in total bacterial population in the bronchoalveolar lavage fluid | 12 weeks
Change in bacterial diversity using Shannon Index based on 16S sequencing. | 12 weeks

SECONDARY OUTCOMES:
Change in bacterial membership using Beta-diversity | 12 weeks
Characterization of bacteria Operational Taxonomic Unit | 12 weeks
Change in total cell count in bronchoalveolar lavage fluid | 12 weeks
Change in total neutrophil count in bronchoalveolar lavage fluid | 12 weeks
Change in total lymphocyte count in bronchoalveolar lavage fluid | 12 weeks
Change in total mono-macrophage count in bronchoalveolar lavage fluid | 12 weeks
Change in St. George's Respiratory Questionnaire | 12 weeks
Change in forced expiratory volume in 1 second | 12 weeks
Change in forced vital capacity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Don Sin, MD, Principal Investigator — St. Paul's Hospital
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho CG, Milne S, Li X, Yang CX, Leitao Filho FS, Cheung CY, Yang JSW, Hernandez Cordero AI, Yang CWT, Shaipanich T, van Eeden SF, Leung JM, Lam S, Sin DD. Airway Eosinophilia on Bronchoalveolar Lavage and the Risk of Exacerbations in COPD. Biomedicines. 2022 Jun 15;10(6):1412. doi: 10.3390/biomedicines10061412. PMID 35740433
- [Derived] Akata K, Leung JM, Yamasaki K, Leitao Filho FS, Yang J, Xi Yang C, Takiguchi H, Shaipanich T, Sahin B, Whalen BA, Yang CWT, Sin DD, van Eeden SF. Altered Polarization and Impaired Phagocytic Activity of Lung Macrophages in People With Human Immunodeficiency Virus and Chronic Obstructive Pulmonary Disease. J Infect Dis. 2022 Mar 2;225(5):862-867. doi: 10.1093/infdis/jiab506. PMID 34610114
- [Derived] Leitao Filho FS, Takiguchi H, Akata K, Ra SW, Moon JY, Kim HK, Cho Y, Yamasaki K, Milne S, Yang J, Yang CWT, Li X, Nislow C, van Eeden SF, Shaipanich T, Lam S, Leung JM, Sin DD. Effects of Inhaled Corticosteroid/Long-Acting beta2-Agonist Combination on the Airway Microbiome of Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Clinical Trial (DISARM). Am J Respir Crit Care Med. 2021 Nov 15;204(10):1143-1152. doi: 10.1164/rccm.202102-0289OC. PMID 34464242